CLINICAL TRIAL: NCT05105633
Title: Extending the Time Window for Tenecteplase by Effective RecanalizatioN of bAsilar Artery occLusion in Patients With POSTerior Circulation Stroke (POST-ETERNAL)
Brief Title: Extending the Time Window for Tenecteplase by Recanalization of Basilar Artery Occlusion in Posterior Circulation Stroke
Acronym: POST-ETERNAL
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT21028
Record Dates: First submitted 2021-10-21; First posted 2021-11-03 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Basilar Artery Occlusion
Keywords: ischemic stroke; basilar artery occlusion; Stroke; Tenecteplase; Tissue Plasminogen Activator; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Fibrin Modulating Agents; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Ischemic Stroke; Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Tenecteplase; Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will receive either intravenous tenecteplase (0.25mg/kg, maximum 25mg, administered as a bolus over 5-10 seconds) or standard of care (alteplase 0.9mg/kg or no lysis) +/- mechanical thrombectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous tenecteplase (TNK) (Experimental): Patients will receive intravenous tenecteplase (0.25mg/kg, maximum 25mg, administered as a bolus over 5-10 seconds).
  Interventions: Drug: Tenecteplase
- Standard Care (which may include intravenous Alteplase) (Active Comparator): Patients will receive standard of care (no intravenous thrombolytic treatment or intravenous alteplase 0.9mg/kg at the standard licensed dose of 0.9 mg/kg up to a maximum of 90mg, 10% as a bolus and the remainder as an infusion over 1 hour).
  Interventions: Drug: Standard Care (which may include intravenous Alteplase)

INTERVENTIONS:
Drug: Tenecteplase — Genetically modified tissue plasminogen activator at a dose of 0.25mg/kg given as an intravenous bolus over 5-10 seconds.
  Arms: Intravenous tenecteplase (TNK)
Drug: Standard Care (which may include intravenous Alteplase) — Patients will receive standard care which may include intravenous alteplase at the standard licensed dose of 0.9 mg/kg up to a maximum of 90mg, 10% as a bolus and the remainder as an infusion over 1 hour.
  Arms: Standard Care (which may include intravenous Alteplase)

SUMMARY:
Patients presenting to the emergency department with an acute ischemic stroke due to basilar artery occlusion within 24 hours of stroke onset will be assessed to determine their eligibility for randomization into the trial. If the patient gives informed consent they will be randomised 50:50 using a central computerised allocation process to either standard of care (no intravenous thrombolytic treatment or intravenous alteplase 0.9mg/kg) or tenecteplase 0.25mg/kg before undergoing mechanical thrombectomy as required at treating clinician's discretion. The trial is Multi-arm, Multi-stage, prospective, randomised, open-label, blinded endpoint (PROBE) design with seamless phase 2b/3 transition if the intermediate endpoint (recanalization without symptomatic intracerebral hemorrhage) is met in analysis of the first 202 patients. Adaptive sample size re-estimation (Mehta and Pocock) will be performed when 240 patients have completed 3 month follow-up (minimum sample size 320, maximum sample size 688).

DETAILED DESCRIPTION:
The study is a Multi-Arm Multi-Stage (MAMS), multiregional, multicentre, prospective, randomised, open-label, blinded endpoint (PROBE), controlled seamless phase 2b/3 trial (2 arm with 1:1 randomisation) with adaptive sample size recalculation in patients with stroke due to basilar artery occlusion. Stage 1 will use the surrogate outcome of recanalization without symptomatic intracerebral hemorrhage (sICH) to establish whether proceeding to Stage 2 is warranted. If results in the first n= 202 patients meet success criteria, the trial will seamlessly convert to a phase 3 design using modified Rankin scale 0-1 at 3 months as the primary outcome (minimum n=320 with interim sample size re-estimation at n=240, maximum sample n=688) using the Mehta and Pocock conditional power method. Each regionally-based stratum will be pooled in the final analysis and analysed as a stratification by geographic region. Randomisation of patients within each stratum will be stratified by the investigator's intention to treat with mechanical thrombectomy (or not) and the investigator's intention to treat with alteplase intravenous thrombolysis should the patient be randomised to the control group (or not). Covariate adjusted minimum sufficient balance randomisation will then be applied to control for age, NIHSS and time from onset-to-randomisation (dichotomized as 0-6 hours vs 6-24 hours). The primary objective of the study is to test the hypothesis that the thrombolytic tenecteplase (TNK, 0.25mg/kg) ± mechanical thrombectomy administered within 24 hours after symptoms onset, is superior to current best practice (alteplase, rtPA, 0.9mg/kg or standard care/no lysis ± mechanical thrombectomy) in achieving excellent functional outcome (mRS 0-1) or return to the premorbid modified Rankin Scale at 90 days in patients with acute ischemic stroke due to basilar artery occlusion. Estimated study duration is 5 years. Patients will participate in the trial for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with posterior circulation ischemic stroke symptoms due to partial or complete basilar artery occlusion within 24 hours from symptom onset (or clinical deterioration/coma) or the time the patient was last known to be well.
* Patient's age is ≥18 years
* Presence of basilar artery occlusion, proven by CT Angiography or MR Angiography. Basilar artery occlusion is defined as 'potentially retrievable' occlusion at the basilar artery. This can be a partial or complete occlusion.
* Premorbid mRS ≤3 (independent function or requiring only minor domestic assistance and able to manage alone for at least 1 week).
* Local legal requirements for consent have been satisfied.

Exclusion Criteria:

* Intracerebral hemorrhage (ICH) or other diagnosis (e.g. tumour) identified by baseline imaging.
* Posterior circulation Acute Stroke Prognosis Early CT score (pc-ASPECTS) <7 on non-contrast CT, CT Angiography source images or DWI MRI.
* Significant cerebellar mass effect or acute hydrocephalus.
* Established frank hypodensity on non-contrast CT indicating subacute infarction.
* Bilateral extensive brainstem ischemia.
* Strong suspicion of underlying intracranial atherosclerotic disease (e.g diffuse arterial calcifications, basilar stenosis) or dissection which may require immediate neuro-interventional procedure with intracranial stenting and not benefit from intravenous thrombolysis at investigator's discretion.
* Pre-stroke mRS of ≥4 (indicating moderate to severe previous disability).
* Other standard contraindications to intravenous thrombolysis.
* Contraindication to imaging with contrast agents.
* Clinically evident pregnant women.
* Current participation in another research drug treatment protocol.
* Known terminal illness such that the patients would not be expected to survive a year.
* Planned withdrawal of care or comfort care measures.
* Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) 0-1 or return to baseline mRS at 90 days | 90 days
  Modified Rankin Scale (mRS) 0-1 (no disability) or return to baseline mRS (if baseline premorbid mRS 2-3) at 90 days

SECONDARY OUTCOMES:
Modified Rankin Scale 0-2 or return to baseline mRS at 90 days | 90 days
  Proportion of patients with Modified Rankin Scale 0-2 or return to baseline mRS at 90 days
Modified Rankin Scale 0-3 or return to baseline mRS at 90 days | 90 days
  Proportion of patients with Modified Rankin Scale 0-3 or return to baseline mRS at 90 days
Ordinal analysis of the mRS at 90 days | 90 days
  Ordinal analysis of the mRS, merging category 5-6, at 90 days
Early clinical improvement | 72 hours
  Proportion of patients achieving early clinical improvement (reduction in acute - 72 hour NIHSS score of ≥8 or 72 hour NIHSS 0-1).
Substantial reperfusion on initial digital subtraction angiography run prior to thrombectomy | Initial angiogram (day 0)
  Proportion of patients with complete occlusion at baseline who achieve eTICI 2b/3 on initial digital subtraction angiography run prior to thrombectomy.
Quality of Life assessment (EQ-5D) - at 90 days and 12 months | 90 days and 12 months
  Quality of Life assessment (EQ-5D) - at 90 days and 12 months
Symptomatic intracerebral hemorrhage (sICH) | 36 hours
  Proportion of patients with sICH defined as parenchymal hemorrhage type 2 (PH2), subarachnoid hemorrhage, and/or intraventricular hemorrhage within 36 of treatment, combined with a neurological deterioration of ≥4 points on the NIHSS from baseline, or leading to death.
All-cause mortality within 90 days | 90 days
  All-cause mortality within 90 days
Modified Rankin Scale (mRS) 5-6 at 90 days | 90 days
  Proportion of patients with Modified Rankin Scale (mRS) 5-6 at 90 days (severe disability or death)

OTHER OUTCOMES:
Intermediate outcome (Stage 1): Partial or complete recanalization of the basilar artery without sICH | Initial angiogram (day 0)
  Proportion of patients achieving partial or complete recanalization of the basilar artery on initial digital subtraction angiography (DSA) prior to thrombectomy or repeat CT Angiography (if DSA not performed) without symptomatic intracerebral hemorrhage (sICH). Partial or complete recanalization is defined as reperfusion of ≥50% of the affected territory or absence of retrievable thrombus.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Campbell, Principal Investigator — University of Melbourne; Fana Alemseged, Principal Investigator — University of Melbourne
Locations (13):
- Australia (13):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Gold Coast Hospital, Gold Coast, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Alfred Health, Melbourne, Victoria
  - Austin Hospital, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
  - Monash Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Western Health, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient data will be uploaded to the Virtual Stroke Trials Archive 2 years after the publication of the primary manuscript. Qualified investigators can access data after submission of a project proposal that has been approved by the VISTA steering committee.
Time Frame: 2 years after the publication of the primary manuscript.
Access Criteria: Qualified investigators can access data after submission of a project proposal that has been approved by the VISTA steering committee.
URL: https://www.virtualtrialsarchives.org/vista/